CLINICAL TRIAL: NCT06002555
Title: A Randomized Open-label, Single Dose, 3-Period, 6-Sequence, Cross-Over Trial With Washout Periods of at Least 14 Days to Investigate the Relative Bioavailability of Apraglutide in Dual Chamber Syringes Versus the Reference Formulation in Vials Following Subcutaneous Administrations in Healthy Subjects
Brief Title: Relative Bioavailability of a New Presentation of Apraglutide Versus the Reference Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VectivBio AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TA799-018
Record Dates: First submitted 2023-07-11; First posted 2023-08-21 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-01

CONDITIONS: Healthy Subjects
Keywords: Relative bioavailability; Dual-chamber syringe
MeSH Terms: interventions — apraglutide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Single SC dose of 5 mg from DCS (Experimental)
  Interventions: Drug: Apraglutide
- Two concomitant single SC doses of 2.5 mg from DCS (Experimental)
  Interventions: Drug: Apraglutide
- Single SC dose of 5 mg from vial (Active Comparator)
  Interventions: Drug: Apraglutide

INTERVENTIONS:
Drug: Apraglutide — Peptide analogue of GLP-2

SUMMARY:
This trial compares the relative bioavailability of apraglutide in dual-chamber syringes (DCS) versus the reference formulation apraglutide in vials.

DETAILED DESCRIPTION:
This is a single-center, open-label, randomized, three-period, and six-sequence cross-over trial with two washout periods of at least 14 days to compare the relative bioavailability of apraglutide using DCS versus the reference formulation in vials, following SC administrations in healthy male and female subjects.

Following consent, subjects will undergo a Screening procedure to see if they are suitable to be enrolled in the trial. Screening may be performed up to 28 days prior to the first injection procedure. All eligible subjects will receive the following treatments in three separate treatment periods:

* Treatment A: Single SC dose of 5 mg (400 µL) from DCS at a concentration of 12.5 mg/mL
* Treatment B: Two concomitant single SC doses of 2.5 mg (400 µL each) of DCS at a concentration of 6.25 mg/mL
* Treatment C: Single SC dose of 5 mg (200 µL) from vial at a concentration of 25 mg/mL of the current formulation-reference There will be a 14-day washout period between the first and second treatment periods and between the second and third treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 67 years inclusive
* Subjects willing and able to comply with the study procedures
* Subjects able to understand and willing to sign the informed consent
* Body mass index (BMI) of ≥18.0 to ≤35.0 kg/m2; and a total body weight of >50 kg
* Women of childbearing potential (WOCBP) having undergone bilateral tubal occlusion or with vasectomized partner. Sterilized or infertile or postmenopausal females.
* Male subjects with a WOCBP partner using highly effective methods of contraception and agreeing on no sperm donation during the trial and for 4 weeks after (EOT) visit.

Exclusion Criteria:

* History of clinically significant gastrointestinal, bronchopulmonary, neurological, cardiovascular, endocrine, or allergic disease
* Known hypersensitivity to the investigational medicinal products (IMP), any of their excipients or drugs of the same class
* If capable of reproduction, unwilling to use an effective form of contraception
* If a WOCBP, a positive blood pregnancy test
* Breast-feeding women
* Positive urine/blood test for alcohol and drugs of abuse
* Use of prohibited medications or herbal remedies
* Known presence or history of intestinal polyps
* Known presence or history of any type of cancer
* Pancreatic events such as acute pancreatitis, pancreatic duct stenosis, pancreas infection, and increased blood amylase and lipase (>2.0-5.0× upper limit of normal range) at Screening or on Day -1 of each period
* Participation in an investigational drug or device study within 30 days prior to screening
* Donation of blood over 500 mL within 3 months prior to screening
* Use of tobacco products (i.e., smokes more than 10 cigarettes per day or equivalent)
* Concomitant disease or condition that could interfere with, or for which the treatment of might interfere with, the conduct of the study, or that would, in the opinion of the Investigator, pose an unacceptable risk to the subject in this trial
* Any intercurrent clinically significant illness in the previous 28 days before Day 1 of this study
* Positive blood screen for human immunodeficiency virus (HIV) antigen/antibody combo, hepatitis A (HAV IGM), hepatitis B surface antigen (HBsAgB), hepatitis B core antigen (anti-HBc) or hepatitis C virus (HCV)
* Unwillingness or inability to comply with the study protocol for any other reason

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Plasma apraglutide primary PK parameter: Maximum observed plasma concentration (Cmax) | 0 to 312 hours post dose in each period
Plasma apraglutide primary PK parameter: AUCinf or AUClast | 0 to 312 hours post dose in each period

SECONDARY OUTCOMES:
Time of maximum plasma concentration (tmax) | 0 to 312 hours post dose in each period
Terminal elimination rate constant (λz) | 0 to 312 hours post dose in each period
Terminal half-life (t½) | 0 to 312 hours post dose in each period
Incidence, nature and severity of adverse events (AE) with apraglutide | Baseline to Day 79
Clinical chemistry | Baseline to Day 79
  Clinical Chemistry panel of analytes will be examined for clinically significant changes.
  Clinical chemistry analytes will be listed by subject. Descriptive statistics will be used to assess any changes in clinical laboratory results during and following trial treatment administration. Values outside the reference ranges will be highlighted and clinical significance stated.
Hematology | Baseline to Day 79
  Hematology panel of analytes will be examined for clinically significant changes.
  Hematology analytes will be listed by subject. Descriptive statistics will be used to assess any changes in clinical laboratory results during and following trial treatment administration. Values outside the reference ranges will be highlighted and clinical significance stated.
Hemostasis | Baseline to Day 79
  Hemostasis INR will be examined for clinically significant changes.
  INR levels will be listed by subject. Descriptive statistics will be used to assess any changes in hemostasis results during and following trial treatment administration. Values outside the reference ranges will be highlighted and clinical significance stated.
Anti-drug antibodies (ADA) analysis | Baseline to Day 79
  ADA will be will be examined for clinically significant changes
Urine analysis | Baseline to Day 79
  Urine analysis panel of analytes will be examined for clinically significant changes.
  Urine analysis data will be listed by subject. Descriptive statistics will be used to assess any changes in clinical laboratory results during and following trial treatment administration. Values outside the reference ranges will be highlighted and clinical significance stated.
Occurrence of clinically relevant changes in electrocardiogram | Baseline to Day 79
  ECG QT Interval
Occurrence of clinically relevant changes in electrocardiogram | Baseline to Day 79
  ECG PR interval
Occurrence of clinically relevant changes in electrocardiogram | Baseline to Day 79
  ECG QRS interval
Occurrence of clinically relevant changes in electrocardiogram | Baseline to Day 79
  ECG rhythm

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Masior, Study Director — VectivBio AG
Locations (1):
- ICON Clinical Research Unit, Groningen, Netherlands